CLINICAL TRIAL: NCT00926250
Title: Effects of Pro-Stat Immuno-Protein Complex (PS-IPC) Supplementation on Muscle Mass and Function, Inflammatory Markers, and Immune Function in Older Adults
Brief Title: Effects of PS-IPC Supplementation on Muscle Mass and Functional Outcomes in Older Adults
Acronym: PS-IPC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor changed their study product and halted study.
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 109167
Record Dates: First submitted 2009-06-22; First posted 2009-06-23 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Immune Senescence; Sarcopenia
Keywords: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PS-IPC supplementation (Experimental)
  Interventions: Dietary Supplement: Oral PS-IPC supplement
- Placebo supplementation (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo supplement

INTERVENTIONS:
Dietary Supplement: Oral PS-IPC supplement — Each subject in this study will be provided the PS-IPC dietary supplement or placebo to consume three times per day for the 12-week duration of the intervention. The placebo supplement will consist of an iso-caloric supplement designed to match the PS-IPC supplement in volume, color, consistency, and palatability.
  Arms: PS-IPC supplementation
Dietary Supplement: Placebo supplement — Each subject in this study will be provided the PS-IPC dietary supplement or placebo to consume three times per day for the 12-week duration of the intervention. The placebo supplement will consist of an iso-caloric supplement designed to match the PS-IPC supplement in volume, color, consistency, and palatability.
  Arms: Placebo supplementation

SUMMARY:
Sarcopenia, the age-associated loss of skeletal muscle mass and strength, is a frequent precursor to functional impairment, disability, falls, and loss of independence in the elderly. The prevalence of sarcopenia is high, with ≥ 45% of the U.S. population aged 60 years or older sarcopenic. Some possible causative factors include a decline in muscle protein synthesis, inactivity, hormonal changes, pro-inflammatory conditions, and reactive oxygen species within the muscle mitochondria, which may all be exacerbated by inadequate nutritional intake. Since dietary protein is targeted to muscle and muscle mass represents the largest tissue in the body, protein nutrition plays a significant role in muscle metabolism.

SPECIFIC AIMS The specific aim of this proposed study is to determine the effect of PS-IPC supplementation on muscle mass, muscle strength, muscle quality, and inflammatory / immune markers in healthy older adults. Subjects scoring 4 - 10 on the Short-Physical Performance Battery and aged 60-85 years will consume PS-IPC supplements or placebo three times daily for 12 weeks.

HYPOTHESES

1. Subjects consuming PS-IPC will have a greater increase in muscle mass and muscle strength compared to a control group consuming a placebo supplement.
2. Subjects consuming PS-IPC will demonstrate a greater increase in the fractional rate of muscle protein synthesis compared with a placebo control group.
3. Subjects receiving PS-IPC will have a reduction in plasma concentrations of various inflammatory markers of immune function, compared to subjects consuming the placebo.

ELIGIBILITY:
Inclusion Criteria:

* BMI of less than or equal to 35 kg/m2, be weight stable (+/- 5 kg) over the previous 4 months (via oral report), report the absence of alcohol or drug abuse, require minimal help in performing activities of daily living, and have a Short Physical Performance Battery score of 4 - 10.

Exclusion Criteria:

* Subjects with acute or chronic disease or who may be using drugs that might interfere with skeletal muscle metabolism / function or immune function will be excluded from participation. Other exclusion criteria include cognitive deficits identified by a Mini-Mental State Examination score < 24, mobility impairment requiring a wheelchair, infections, endocrine diseases (e.g., diabetes or untreated thyroid dysfunction), active inflammatory conditions, autoimmune disorders, renal dysfunction, anemia (hemoglobin < 11.5 g/dL), cardiac problems in preceding 3 months or congestive heart failure, chronic obstructive lung disease, neoplasia other than of the skin during the preceding 5 years, influenza vaccine within last 3 weeks or other vaccines within last 6 weeks, known systemic reaction to any immune function test antigen, and use of the following drugs: immunosuppressants, antianginal agents, antiarrhythmics, antibiotics within last 2 weeks, and oral steroids. Other conditions may be used as inclusion / exclusion criteria at the discretion of the study physician to ensure the safe participation of potential study subjects.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Muscle protein synthesis | 14-16 months

SECONDARY OUTCOMES:
Body composition | 14-16 months
Skeletal muscle strength and function | 14-16 months
Immune function | 14-16 months
Physical activity level | 14-16 months
Self-perceived quality of life | 14-16 months

CONTACTS AND LOCATIONS:
Overall Officials: Arny A Ferrando, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States